CLINICAL TRIAL: NCT05258734
Title: The Effect Of Mobile Health Application Based On Omaha System On Physical, Psychosocial, Cognitive Symptoms And Quality Of Life In COVID-19 Patients
Brief Title: The Effect of Mobile Health Application Based on Omaha System on Symptoms and Quality of Life in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gizemnur Torun, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4802180417
Record Dates: First submitted 2022-02-05; First posted 2022-02-28 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Symptoms and Signs; Quality of Life
Keywords: Omaha System; Mobile health app
MeSH Terms: conditions — COVID-19; Signs and Symptoms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVOS app (Experimental)
  Interventions: Other: COVOS app
- Control Group (Active Comparator)
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: COVOS app — In this study, the patients in the experimental group will be followed up with the COVOS app and nursing interventions (videos, information messages) to manage their symptoms will be directed with the COVOS app.
  Arms: COVOS app
Other: Standard Care — In this study, the patients in the control group will not receive any intervention, the standard follow-up and health care provided by the family health center of the patients will continue.
  Arms: Control Group

SUMMARY:
Purpose: The aim of this study is to evaluate the effects of nursing interventions made with a mobile health application (COVOS) developed based on the Omaha System on the physical, psychosocial and cognitive symptoms and quality of life of patients diagnosed with COVID-19, and continuing treatment at home.

Design: This is a single center, 1:1 randomized, single blind, parallel, active comparator trial.

Method: Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) Statement 2013 checklist used in study. The CONSORT (Consolidated Standards of Reporting Trials) flowchart is used in this protocol. This study will carried out in a family health center, located within the boundaries of İzmit District of Kocaeli province. The patients in the experimental group will be followed up with the COVOS app and nursing interventions (videos, information messages) to manage their symptoms will be directed with the COVOS app. The patients in the control group will not receive any intervention, the standard follow-up and health care provided by the family health center of the patients will continue.

Hypothesis: In patients diagnosed with COVID-19 followed at home with COVOS, symptom management and quality of life will be better in 1st, 2nd and 3rd months compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a positive Polymerase Chain Reaction (PCR) test within the last 24-48 hours
* Patients whose symptoms started within the last 48 hours
* Patients experiencing at least one symptom
* Patients diagnosed with COVID-19 and continuing treatment at home
* Literate patients
* Patients with smartphone

Exclusion Criteria:

* Those who have had a previous COVID-19 infection
* Patients with vision or hearing problems
* Patients with chronic disease
* Patients with mental illness
* Patients who do not have a smartphone
* Pregnant and postpartum patients
* Patients who did not agree to participate in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-23 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Change in Physical Symptom Status | Baseline, 1st month, 2nd month and 3rd month.
  Physical symptom status will be assessed using the Omaha System Problem Rating Scale for Outcomes. The Problem Rating Scale for Outcomes is a method to evaluate patient progress throughout the period of service. It consists of three five-point, Likert-type scales to measure the entire range of severity for the concepts of Knowledge, Behavior, and Status.
Change in Psychosocial Symptom Status | Baseline, 1st month, 2nd month and 3rd month.
  Psychosocial symptom status will be evaluated with Depression Anxiety Stress Scale- 21 (DASS-21). DASS-21 is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. For depression the cutoff scores are: Normal: 0-9, Mild: 10-12, Moderate:13-20, Severe: 21-27, and Extremely severe: 28-42.
  For anxiety the cutoff scores are: Normal: 0-6, Mild: 7-9, Moderate: 10-14, Severe:15-19, and Extremely severe: 20-42. For stress the cutoff scores are: Normal: 0-10, Mild:11-18, Moderate:19-26, Severe: 27-34, and Extremely severe: 35-42.
Change in Cognitive Symptom Status | Baseline, 1st month, 2nd month and 3rd month.
  Cognitive symptom status will be assessed using the Omaha System Problem Rating Scale for Outcomes. The Problem Rating Scale for Outcomes is a method to evaluate patient progress throughout the period of service. It consists of three five-point, Likert-type scales to measure the entire range of severity for the concepts of Knowledge, Behavior, and Status.
Change in Quality of Life | Baseline, 1st month, 2nd month and 3rd month.
  Quality of life will be evaluated with the SF-12. The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
  The SF-12 uses the same eight domains as the SF-36:
  Limitations in physical activities because of health problems. Limitations in social activities because of physical or emotional problems Limitations in usual role activities because of physical health problems Bodily pain General mental health (psychological distress and well-being) Limitations in usual role activities because of emotional problems Vitality (energy and fatigue) General health perceptions

CONTACTS AND LOCATIONS:
Overall Officials: Selda Seçginli, Prof.Dr., Study Director — İstanbul University Cerrahpasa
Locations (1):
- Kocaeli University, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No